CLINICAL TRIAL: NCT00855985
Title: A Randomised Controlled Trial of Pancreaticogastrostomy Versus Pancreaticojejunostomy in Reconstruction After Pancreaticoduodenectomy for Cancer
Brief Title: Anastomotic Techniques in Pancreaticoduodenectomy
Acronym: PG/PJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lakeshore Hospital (Other)
Responsible Party: Principal Investigator, Dr H Ramesh, Director of Surgical Gastroenterology, Lakeshore Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Pancreatic Cancer; Pancreatic Fistula
Keywords: Pancreatic anastomosis; Whipple operation
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pancreaticojejunostomy for reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: type of anastomosis after pancreaticoduodenectomy
- 2 (Active Comparator): Pancreaticogastrostomy for reconstruction after pancreaticoduodenectomy
  Interventions: Procedure: type of anastomosis after pancreaticoduodenectomy

INTERVENTIONS:
Procedure: type of anastomosis after pancreaticoduodenectomy — pancreaticojejunostomy (arm 1) versus pancreaticogastrostomy (arm 2)for reconstruction of the pancreatic remnant after pancreaticoduodenectomy

SUMMARY:
There are two principal ways of draining the remnant of the pancreas back into the intestine after removal of the head of the pancreas for cancer. This can be performed either to the jejunum or to the stomach. The aim of this study is to randomly allocate consenting patients to one of the two arms to study whether the leak rates from the anastomosis and the outcomes after the surgery are affected.

Previous papers have shown similar results in both groups although non randomized data suggested that the Pancreaticogastrostomy (drainage into the stomach) may be superior

ELIGIBILITY:
Inclusion Criteria:

1. Pancreaticoduodenectomy for adenocarcinoma of the pancreatic head
2. resectable tumour

Exclusion Criteria:

1. chronic pancreatitis/benign tumours-
2. tumours extending into the body of the pancreas
3. tumours with metastasis beyond regional lymph nodes
4. requirement for sub total pancreatectomy
5. prolonged hypotension - < 80 mm of hg for more than 30 min

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2004-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula rate | 30 days

SECONDARY OUTCOMES:
mortality | 90 days
Hospital stay | 90 days
need for postoperative intervention | 90 days
major complication | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Hariharan Ramesh, MS MCh, Principal Investigator — Lakeshore Hospital
Locations (1):
- Lakeshore Hospital & Research Center, Kochi, Kerala, India